CLINICAL TRIAL: NCT05491590
Title: Patient-reported Outcomes in Status Epilepticus Requiring Intensive Care Unit Management
Brief Title: Patient-reported Outcome After Status Epilepticus
Acronym: POSEIDON
Status: Completed | Type: Observational
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Jacq Gwenaelle, Investigator Coordinator, Versailles Hospital
Other Study IDs: P21/11 - POSEIDON
Record Dates: First submitted 2022-08-01; First posted 2022-08-08 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Patient Reported Outcomes; Long Term Outcomes; Status Epilepticus; Intensive Care Unit; Intensive Care Unit Syndrome
MeSH Terms: conditions — Status Epilepticus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Status epilepticus (SE) is a common life-threatening neurological emergency in which prolonged or multiple closely spaced seizures can result in long-term impairments. SE remains associated with considerable mortality and morbidity, with little progress over the last three decades. The proportion of patients who die in the hospital is about 20% overall and 40% in patients with refractory SE. Morbidity is more difficult to evaluate, as adverse effects of SE are often difficult to differentiate from those attributed to the cause of SE. Our experience suggests that nearly 50% of patients may experience long-term functional impairments.

The precise description of the consequences of these functional impairments and their impact on quality of life after SE requiring intensive care management has been little studied.

Indeed, if cognitive, physical and mental impairments are now identified in the populations of patients who required intensive care under the term post-resuscitation syndrome (PICS), neuronal lesions consecutive to the SE itself or to its cause could be responsible for these different functional alterations. Thus, the following have been described: (i) cognitive disorders in the areas of attention, executive functions and verbal fluency, visual and working memory disorders, but also spatio-temporal disorders; (ii) physical disorders such as the so-called post-resuscitation polyneuromyopathy; and (iii) mental disorders such as anxiety disorders, depressive states or those related to post-traumatic stress.

Assessment and characterization of patient-reported outcomes is essential to complement the holistic assessment of clinically relevant outcomes from the patient's perspective. Here, we propose the development of a cross-sectional collection of PROs of the different constituents of PICs and HR-QOLs, and associated with functional patient outcomes, in those who required ICU management for status epilepticus.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years old or older
* Patients previously included in the ICTAL registry (Status Epilepticus cohort NCT03457831)
* Survivors after ICU management for Status Epilepticus More than 3 months and less than 5 years after ICU discharge

Exclusion Criteria:

* Legal guardianship
* Opposition to participate
* Unread and unwritten French language
* Patient not affiliated to a Social Security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who meet the eligibility criteria will be offered participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
percentage of global impairment of HRQoL defined by one and/or other of the physical and mental impairments (after dichotomization of the SF 36 summary scores compared to the general population) in patients managed in the ICU for or with SE. | one day
  36-Item Short Form Survey (SF-36) (HRQoL)-Ranging score[0-100], a high score indicate better health status.

SECONDARY OUTCOMES:
percentage of cognitive/physical and/or mental health impairment defined after dichotomization of i)T-MoCA ,ii) GOS, iii)IADL&ADL, iv)HAD, v)IES-r in patients managed in the ICU for or with SE | one day
  * i)The Montreal Cognitive Assessment (MoCA)(Cognition)-Ranging score[0-30] a score of 26 and higher generally is considerednormal or Telephone MoCA-Ranging score[0-22],a score of 18 and higher generally is considered normal.
  * ii)The Glasgow Outcome Scale extended (Handicap)-Ranging score[1-8] a hight score indicate no handicap
  * iii) The Lawton IADL (scale contains eight items, with a summary score from 0 (low function) to 8 (high function). Each ability measured by the scale relies on either cognitive or physical function, though all require some degree of both.
  * and Barthel index (Dependency)-Ranging score[0-100], a high score indicate no dependency.
  * iv)The Hospital anxiety and depression (Anxiety,Depression)-Ranging score[0-21] a score > 8 indicate in each subscale a depresion or/and anxiety
  * v)The Impact of Event Scale -Revised(post traumatic syndrome disorder)-Ranging score[0-88],scores higher than 24 are of concern; the higher scores indicate the severity of PTSD
percentage of impairement of HRQoL, in 8 dimensions of the generalist of SF 36, and scores in the 7 dimensions of the specific QOLIE 31 in patients managed in intensive care for or with SE. | one day
  -QOLIE 31 measure of spécific QoL of epileptics patients, 30 items are organized into seven subscales:Ranging score[0-100], a high score indicate better health status.
percentage of impairement of HRQoL, in 8 dimensions of the generalist of SF 36, and scores in the 7 dimensions of the specific QOLIE 31in the SE sub-groups defining (with or without predominant motor signs) | one day
  * 36-Item Short Form Survey (SF-36) (HRQoL)-Ranging score[0-100], a high score indicate better health status.
  * QOLIE 31 measure of spécific QoL of epileptics patients, 30 items are organized into seven subscales:Ranging score[0-100], a high score indicate better health status.
Presence or absence Post-ICU factors associed to the PICs, as defined above in patients managed in the ICU for or with SE. | one day
  cf outcomes 2
Presence or absence of the elements associated with the PICs, as defined above, in the subgroups defining SE (SE with orwithout predominant motor signs,). | one day
  * i)The Montreal Cognitive Assessment (MoCA)(Cognition)-Ranging score[0-30] a score of 26 and higher generally is considerednormal or Telephone MoCA-Ranging score[0-22],a score of 18 and higher generally is considered normal.
  * ii)The Glasgow Outcome Scale extended (Handicap)-Ranging score[1-8] a hight score indicate no handicap
  * iii) The Lawton IADL (scale contains eight items, with a summary score from 0 (low function) to 8 (high function). Each ability measured by the scale relies on either cognitive or physical function, though all require some degree of both.
  * and Barthel index (Dependency)-Ranging score[0-100], a high score indicate no dependency.
  * iv)The Hospital anxiety and depression (Anxiety,Depression)-Ranging score[0-21] a score > 8 indicate in each subscale a depresion or/and anxiety
  * v)The Impact of Event Scale -Revised(post traumatic syndrome disorder)-Ranging score[0-88],scores higher than 24 are of concern; the higher scores indicate the severity of PTSD
Presence or absence Post-ICU factors associated of return to work ability in patients managed in the ICU for or with SE. | one day
  A return to work or school will be interpreted by the structured GOS interview.
score of perceived social support by the SSQ6 scale in its 2 dimensions, satisfaction and availability. | one day
  The Social Support Questionnaire- Short Form-SSQ6 / 6 item measure of social support, with scores ranging from 0 (no social support) to 6 (very high social) and 1 (very dissatisfied) to 6 (very satisfied) for the area of satisfaction in each item or area. From these scores in the 6 domains, an average score was calculated for the number of supports available -Ranging score[0-54] and for satisfaction.Ranging score[0-36]
percentage of the quality of life impairement in the total population and in in the SE sub-groups patients identified with an previous epilepsy | one day
  * 36-Item Short Form Survey (SF-36) (HRQoL)-Ranging score[0-100], a high score indicate better health status.
  * QOLIE 31 measure of spécific QoL of epileptics patients, 30 items are organized into seven subscales:Ranging score[0-100], a high score indicate better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Gwenaelle JACQ, RN,MSc,PhDc, Principal Investigator — Versailles Hospital; Stephane LEGRIEL, MD,PhD, Study Director — Versailles Hospital
Locations (16):
- France (16):
  - CHVersailles, Le Chesnay, Yvelines
  - CH de Bethune, Beuvry
  - CHU de Brest, Brest
  - CH de Brive la Gaillarde, Brive-la-Gaillarde
  - CH de Cannes, Cannes
  - CH du Cotentin, Cherbourg
  - CHU de Beaujon, Clichy
  - CHU Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - CH de la Rochelle, La Rochelle
  - GH Sud Ile de France, Melun
  - CHU de Nantes, Nantes
  - GH Paris Saint Joseph, Paris
  - Hôpital Claude Galien, Quincy-sous-Sénart
  - CH de Roanne, Roanne
  - CH de Toulon-La Seyne sur Mer, Toulon